CLINICAL TRIAL: NCT01506544
Title: Pharmacokinetics and Relative Bioavailability of a Liquid Formulation of Hydroxyurea in Pediatric Patients With Sickle Cell Anemia
Brief Title: Pharmacokinetics (PK) of Liquid Hydroxyurea in Pediatric Patients With Sickle Cell Anemia
Acronym: HU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kathleen A Neville, Associate Professor of Pediatrics, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: Hydroxyurea Pharmacokenetic; HHSN275201000003I (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2011-09-30; First posted 2012-01-10 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Sickle Cell Anemia
Keywords: HU; Hydroxyurea; Sickle cell; Pediatric
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 Pharmacokinetic study (Experimental): This will be a single dose study where participants will receive 20mg/kg or the participant's usual dose as a liquid containing hydroxyurea 100mg/mL. For a subset of participants (n= at least 6), a multiple-dose, steady state (i.e. at least 4 consecutive days of dosing) study will be performed.
  Interventions: Drug: Hydroxyurea
- Arm 2: Relative bioavailability study (Active Comparator): This will be a single dose study. Participants will receive each of the two following treatments of HU in a randomized, crossover fashion: Either approximately 20 mg/kg/day (rounded to the nearest 200mg and no greater than 30 mg/kg) or the participant's usual daily dose as: 1) a liquid containing 100 mg/mL of hydroxyurea, or 2) Droxia® 200 mg capsules administered orally.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — 20mg/kg of Hydroxyurea or the patient's standard daily dose
  Other Names: Droxia Capsules; Hydrea

SUMMARY:
Hydroxyurea (HU) is approved by the United States Food and Drug Administration (FDA) to treat adults with sickle cell anemia. Hydroxyurea has also been tested and used with children with sickle cell anemia. However, there are not many studies describing the disposition of drug in children less than 5 years old. The FDA has requested this study to better understand how children ages 2 to 17 years with sickle anemia absorb and eliminate the drug (this is called pharmacokinetics). The investigators will measure how much Hydroxyurea (HU) gets into the bloodstream at different time points after taking this medication.

ELIGIBILITY:
For Both Arms:

Pharmacokinetics and Relative Bioavailability of a Liquid Formulation of Hydroxyurea in Pediatric Patients with Sickle Cell

* The study participant will be a pediatric (male or female) participant with sickle cell anemia with laboratory (i.e. electrophoretic, chromatographic or DNA) confirmation of the diagnosis of Hemoglobin SS or Sβ0thalassemia.
* Weight ≥ 10 kg.
* Participants may or may not be currently receiving hydroxyurea. If participants are taking hydroxyurea, the last dose must be no less than 24 hours prior to the start of the study.
* Participant is in the "well" state (i.e. at least 2 weeks since the last vaso-occlusive crisis, acute chest syndrome episode, or splenic sequestration episode).
* Clinical evidence of normal gastrointestinal function and structure.
* No clinical evidence of hepatic compromise including transaminases no more than 3 times the upper limit of normal.
* A glomerular filtration rate (GFR--estimated from serum creatinine using age-appropriate, validated equations such as the Schwartz equation) > 70 ml/min/1.73m2 and no known renal impairment (creatinine no more than 1.5 times the upper limit of normal for age in the screening laboratory).
* Body mass index (BMI) ≥5th and ≤ 95th percentile as per CDC growth charts.
* The parent or guardian is willing and able to provide a signed and dated written informed consent form prior to any study related procedures. When appropriate, the participant has signed an assent to participate according to local IRB guidelines.
* The participants and/or participant's parents are able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions such that the participant is likely to complete the study as planned.
* Based on the opinion of the physicians providing patient care and those conducting the study, there are no apparent contraindications for inclusion as a participant in a pharmacokinetic study.
* For the Pharmacokinetic Study (Arm 1):
* Participant is ≥ 2 years and ≤ 5 years of age.
* The participant is able to consume a minimum of 30 ml of water following ingestion of the study article.
* For the Relative Bioavailability Study:
* Participant is > 5 years and < 17 years of age.
* All females of child-bearing potential must be found to have a negative serum pregnancy test prior to initial dosing and be willing to practice appropriate contraceptive measures, including abstinence, from the time of the initial pregnancy testing through the remainder of the study (30 days after last administration of investigational agents).
* The participant is able to ingest both capsule and liquid study articles and consume a minimum of 30 ml of water following ingestion of medication.

EXCLUSION CRITERIA

* A participant will not be eligible for inclusion in this study if any of the following criteria apply:
* Chronic transfusion therapy, or transfused within 3 months of study participation.
* Known renal impairment (creatinine greater than 1.5 times the upper limit of normal for age in the screening laboratory).
* Known hepatic impairment or elevated transaminases (greater than 3 times normal).
* Known presence of malignancy.
* The participant is unwilling and/or unable to abstain from use of tobacco- or nicotine-containing products for 24 hours prior to screening and for 24 hours prior to dosing until collection of the final PK sample during each treatment period.
* Diagnoses other than sickle cell anemia or sickle beta-zero thalassemia (i.e., other sickle cell variants or sickle hereditary persistence of fetal hemoglobin).
* Blood count parameters as follows: Hemoglobin less than 6.0 gm/dL, absolute reticulocyte count less than 80,000 mm-3, neutrophil count less than 1200 mm-3, platelet count less than 150,000 mm-3.
* The participant has used opiates, H2 blockers, proton pump inhibitors, antacids, other GI motility agents or any other medication that, in the opinion of the investigator and/or sponsor, will interfere with the study procedures or affect the interpretation of the results of the study for 3 days prior to the first dose of study.
* Use of over the counter non-steroidal anti-inflammatory agent or narcotic analgesic within 3 days.
* Participant has received an investigational drug within the past 30 days.
* Use of any illicit or illegal substances.
* The parent or guardian is unwilling or unable to provide a signed and dated written informed consent form prior to any study related procedures, or, when appropriate, the participant has refused to sign an assent to participate according to local IRB guidelines.
* Any other condition or chronic illness, which in the opinion of the Principal Investigator makes participation unadvised or unsafe.
* The caregiver is unwilling or unable to provide a completed study diary for a participant in the steady-state subset.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics | predose, 0.17, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose
  Cmax, Area Under Curve, Tmax. Also, the following pharmacokinetic parameters will be derived for each participant using standard techniques: Apparent absorption rate constant, Apparent terminal elimination rate constant, Apparent steady state volume of distribution, Apparent plasma clearance. A compartment, model-based, classical fitting paradigm of the plasma concentration vs. time data will be applied to each subjects' data. Standard goodness of fit criteria will be employed. Subjects aged greater than or equal to 2 and less than or equal to 17 years.
Pharmacokinetics of HU | predose, 0.17, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose
  To evaluate the relative bioavailability of a liquid HU formulation (100mg/mL0 in participants ages greater that 5 and less than or equal to 17 years of age compared to standard therapy utilizing Droxia 200mg capsules

SECONDARY OUTCOMES:
Bioavailability of HU | predose, 0.17, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8 hours post-dose
  Relative bioavailability of liquid HU formulation in comparison to Droxia® capsules will be assessed according to published FDA Bioequivalence Guidance Subjects aged greater than 5 and less than or equal to 17 years Derived steady-state PK parameters after multiple doses of liquid HU (AUC(0-12), AUC(0-∞), Cmax, Tmax, and t½) Steady-state plasma(PK)parameters for liquid formulation of HU will be evaluated Subjects ages greater than or equal to 2 and less than or equal to 5 years will receive doses of 20mg/kg/day for at least 4 consecutive days before evaluation of the steady-state parameters

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Neville, MD, MS, Principal Investigator — Children's Mercy Hosptials and Clinics
Locations (6):
- United States (6):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Memorial Hospital (Northwestern University), Chicago, Illinois
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - UT Southwestern University Hospital, Dallas, Texas
  - Children's Hospital of Wisconsin, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Estepp JH, Wiczling P, Moen J, Kang G, Mack JM, Liem R, Panepinto JA, Garg U, Kearns G, Neville KA. Hydroxycarbamide in children with sickle cell anaemia after first-dose vs. chronic therapy: pharmacokinetics and predictive models for drug exposure. Br J Clin Pharmacol. 2018 Jul;84(7):1478-1485. doi: 10.1111/bcp.13426. Epub 2017 Nov 28. PMID 28884840